CLINICAL TRIAL: NCT03145324
Title: Immunisation History Survey - a Study to Measure Levels of Immunity to Routine Immunisations
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OVG 2012/08
Record Dates: First submitted 2013-10-16; First posted 2017-05-09 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2017-05

CONDITIONS: Immunization; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Collection of vaccine histories

SUMMARY:
To collect the immunisation history of participants enrolled in a previous vaccine study (REC 09/H0604/107) in order to assess the influence of genetic variation on the level of immunity to routine immunisations.

DETAILED DESCRIPTION:
Children aged 6 month to 13 years were enrolled in a study to compare the immunogenicity and safety of adjuvanted or non-adjuvanted influenza vaccines during the 2009 pandemic influenza season. Nine-hundred and forty-nine children were recruited from 5 UK centres: Oxford, Southampton, Bristol, Exeter, and London

In the previous study, DNA was collected when individuals provided appropriate consent, to explore the genetic determinants of responses to vaccination. Although, study participants consented for their medical records to be reviewed by members of the study team, and for these data as well as anonymised serum samples to be used in future research, routine immunisation histories were not collected before this study closed.

In this study we wish to collect the full vaccination history of participants, as this information will be extremely important in interpreting results. We propose sending a letter to parents/guardians informing them of the study and asking whether they are willing for members of the study team to approach their general practitioner or the child health computer system in order to retrieve these records. Immunisation histories will then be included with other non-identifiable information needed for analysis, and samples unlinked from personal identifiers prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are consent in the original vaccine study (09/H0604/107) with explicit consent for samples to be stored and used in future research as well as consent to this subsequent study

Exclusion Criteria:

* Individuals who do not have explicit consent for samples taken in the original vaccine study (09/H0604/107) to be stored for future research.
* Individuals who have not been consented into this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants enrolled in a previous vaccine study (REC 09/H0604/107)
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the completion of the collection of vaccination histories from consented participants. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard Pollard, PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- See also: Related Info — http://www.ovg.ox.ac.uk/recruiting-studies